CLINICAL TRIAL: NCT04283786
Title: The BLAST OFF (Bisphosphonate aLternAtive regimenS for the prevenTion of Osteoporotic Fragility Fractures) Study
Brief Title: Exploring Efficacy, Cost Effectiveness and Experiences Related to Adherence of Different Bisphosphonate Regimens for the Prevention of Osteoporotic Fragility Fractures.
Acronym: BLASTOFF
Status: Completed | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 43961
Record Dates: First submitted 2020-02-18; First posted 2020-02-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Osteoporosis
Keywords: bisphosphonates; systematic review; qualitative interviews; osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- General Practitioner: General Practitioners working within primary care in the UK
  Interventions: Other: Qualitative Interview
- Primary Care Patients: Patients cared for in primary care who started on oral bisphosphonates within the last 24 months for prevention of fragility fractures
  Interventions: Other: Qualitative Interview
- Secondary Care Clinicians: Clinicians working in secondary care as specialists (e.g. nurses, consultants) involved in the treatment of osteoporosis
  Interventions: Other: Qualitative Interview
- Secondary Care Patients: Patients cared for in secondary care receiving hospital based (intravenous) bisphosphonate treatments for prevention of fragility fractures who began treatment within the last 24 months
  Interventions: Other: Qualitative Interview
- Clinical Academics: Clinical academics involved in osteoporosis research
  Interventions: Other: Qualitative Interview
- Secondary Care Clinicians - Novel Care: Clinicians working in secondary care as specialists (e.g. nurses, consultants) from the osteoporosis service in Nottingham and Sheffield with insight into alternate bisphosphonate treatments
  Interventions: Other: Qualitative Interview
- Secondary Care Patients - Novel Care: Patients cared for in secondary care receiving alternative bisphosphonate treatments for prevention of fragility fractures who began treatment within the last 24 months at the osteoporosis service in Nottingham or Sheffield
  Interventions: Other: Qualitative Interview
- Commissioners: Commissioners involved in osteoporosis services
  Interventions: Other: Qualitative Interview

INTERVENTIONS:
Other: Qualitative Interview — A single qualitative interview about experiences of bisphosphonate regimens, as well as wider experiences of service quality and delivery.

SUMMARY:
Osteoporosis is a condition where bones become weak and fragile and can easily break. Suffering from one fragility fracture doubles your chance of having another. These fractures can affect a person's life significantly and contribute to significant costs to the UK (United Kingdom) health service.

Bisphosphonates are used to treat osteoporosis and help prevent fractures. The most commonly used bisphosphonate treatment is Alendronate, but taking it correctly is complicated and side-effects are common. Therefore only 1 in 4 people continue with Alendronate beyond 2 years. There are different forms of bisphosphonates that can be given in different ways and frequencies and may be more acceptable and tolerated by patients.

The study will look at how effective different bisphosphonate regimens are compared to Alendronate at preventing fractures, whether the reduction in fracture risk can be achieved at reasonable financial cost and establish acceptability of different approaches to patients.

The study will be completed in 2 stages, Stage 1A and Stage 1B in parallel, followed by Stage 2.

Stage 1A will update a systematic review to inform which regimens are most effective at reducing fractures and provide the best value for money.

Stage 1B will consist of qualitative, semi-structured interviews from a sample of stakeholders in receipt of or involved in the delivery of different bisphosphonate regimens, in order to identify which bisphosphonate regimens are most acceptable to patients and the barriers to effective compliance and adherence.

Stage 2 will use focus groups and workshops with stakeholders and commissioners to discuss uncertainties from Stage 1 and identify the most important outstanding questions for future research.

DETAILED DESCRIPTION:
This information provided relates to Stage 1B. Stage 1A does not involve participants. Stage 2 will be conducted by the Royal Osteoporosis Society. Participants will not be invited via NHS (National Health Service) organisations and no identifiable information will be collected.

Participants are only involved in Stage 1B of the study, which consists of qualitative interviews only. Participants will be drawn from several different areas of healthcare, in order to ensure a best range of relevant patients', clinicians', commissioners', service managers' and researchers' experiences. Patient participants will be identified as potentially eligible by their healthcare providers, either via their GP (General Practitioner) surgery or secondary care clinician.

Patients will receive a Study Information Pack via the post, containing an Invitation (Patient) Letter from their GP or responsible secondary care doctor, a Participant (Patient) Information Sheet, a reply slip and a freepost envelope with the Research Team's return address. This information pack will also include the Research Team's contact details in order that potential participants have an opportunity to ask questions before indicating an interest in taking part in the study. Patients may also contact the Research Team to express interest by response to a Patient Information Poster in certain service areas, and they will be supplied with the same Study Information Pack. Patients who return a reply slip will be contacted by a member of the Research Team to arrange a convenient time and location in which to obtain written informed consent and undertake the semi-structured interview, which is likely to be immediately after written consent is obtained.

Non-patient participants will be identified as potentially eligible via their General Practice Managers or via snowball sampling from their Service Lead in secondary care services. They will be provided with an Invitation (Clinician) Letter/Email and Participant (Clinician) Information Sheet. The information pack will also include the Research Team's contact details in order that potential participants have an opportunity to ask questions before indicating an interest in taking part in the study. If they indicate to the Research Team they would like to participate in the study, a member of the Research Team will contact the participant to obtain written informed consent, before arranging a convenient time and location to undertake the semi-structured interview, which may be immediately after written consent is obtained.

The semi-structured interviews will be conducted face-to-face or by telephone and are expected to take 40-50 minutes to complete. Face-to-face interviews will be conducted in a private setting either within the site of treatment or at their home in the case of a patient participant, or within the place of work for non-patient participants.

The interview guide will be developed iteratively throughout the study to cover issues as identified from the scoping review of published studies assessing experiences of bisphosphonate regimens, as well as wider experiences of service quality and delivery. This will include questions around patient factors (such as values and health beliefs), service factors (location, accessibility, assurance, and empathy), relational factors (provider patient relations) and medication factors (dosing complexity, frequency, side effects). Clinician interviews will also include barriers to maintain a service around alternative bisphosphonates regimens, as well as changes in service over time.

Interviews will be undertaken by qualitative researchers (employed by University of Nottingham). Interviews will be audio-recorded and then transcribed by Clayton Research Support, a Nottingham University Hospitals and University of Nottingham approved transcription service.

There is no intervention involved in this study. Once the interview is completed, a participant's involvement in the study is ended. There is no further follow-up.

Thematic analysis of interview data will be conducted. This will involve familiarisation, identification of a framework, and interpretation, paying particular attention to themes clustered around service variables. The analysis will involve a preliminary phase of more general qualitative data analysis (close reading of transcripts, open coding, identification of themes). Analysis will be undertaken in the first instance by the Research Fellow alongside and overseen by the Stage 1B Lead. Emerging themes (with all identifying information removed) will be discussed at appropriate intervals with the wider study management group. The approach will allow for both a-priori and emergent codes to be identified. NVivo software will be used to develop an appropriate coding strategy and framework.

Due to the Covid-19 pandemic and the need for a contingency recruitment plan, Non-substantial Amendment 02 was submitted and approved on 15th May 2020 to facilitate patient recruitment from the Royal Osteoporosis Society members via newsletter article, allowing interviews to be conducted by telephone rather than face-to-face at a specific location.

ELIGIBILITY:
Inclusion Criteria:

Adults over the age of 18 with the ability to give informed consent and represent one of the following stakeholder groups:

1. GPs
2. Patients who started on oral bisphosphonates within the last 24 months for prevention of fragility fractures
3. Secondary care specialist clinicians (nurses, consultants) involved in the treatment of osteoporosis.
4. Patients receiving hospital based (intravenous) bisphosphonate treatments for prevention of fragility fractures who began treatment within the last 24 months
5. Clinical academics involved in osteoporosis research
6. Specialist clinicians (nurses, consultants) from the osteoporosis service in Nottingham and Sheffield with insight into alternate bisphosphonate treatments
7. Patients receiving alternate bisphosphonate treatments for prevention of fragility fractures who began treatment within the last 24 months
8. Commissioners involved in osteoporosis services

Exclusion Criteria:

1. Patients who take bisphosphonate medicines for reasons other than osteoporosis or osteopenia, including patients with an active cancer, primary hyperparathyroidism and Paget's disease.
2. Are unable to give informed consent
3. Considered to be near to end of life.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients and stakeholders in receipt of or involved in the delivery of bisphosphonate treatment for the prevention of fragility fractures.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Views, experiences and preferences of patients, clinicians and researchers regarding different bisphosphonate treatment regimens. | 40-50 minutes
  Collected through conduction and analysis of semi-structured interviews.

SECONDARY OUTCOMES:
Effectiveness of different bisphosphonate regimens in preventing fragility fractures in adults. | 24 months
  By analysis of published literature by systematic review.
Cost-effectiveness of different bisphosphonate regimens in preventing fragility fractures in adults. | 24 months
  Using a health economic model on data of published literature identified by systematic review
Prioritised future research questions regarding the effectiveness and adherence profile of different bisphosphonate regimens in preventing fragility fractures in adults. | 2-3 hours
  By stakeholder engagement workshops using the James Lind methodology.

CONTACTS AND LOCATIONS:
Overall Officials: Opinder Sahota, Professor, Principal Investigator — Nottingham University Hospitals NHS Trust
Locations (1):
- Nottingham University Hospitals Trust, Queens Medical Centre, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The datasets (whole transcripts) generated during and/or analysed during the current study are not expected to be made available due to participant confidentiality.
  Some anonymised statements may be available within the published results.